CLINICAL TRIAL: NCT05827016
Title: A Phase 3, Two-stage, Randomized, Multi-center, Controlled, Open-label Study Comparing Iberdomide Maintenance to Lenalidomide Maintenance Therapy After Autologous Stem Cell Transplantation (ASCT) in Participants With Newly Diagnosed Multiple Myeloma (NDMM) (EXCALIBER-Maintenance)
Brief Title: A Study to Compare Iberdomide Maintenance Versus Lenalidomide Maintenance Therapy Following Autologous Stem Cell Transplant in Participants With Newly Diagnosed Multiple Myeloma
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IM048-022; U1111-1280-9492 (Other: WHO); 2022-501515-14-00 (Other: EU CTR)
Record Dates: First submitted 2023-04-11; First posted 2023-04-24 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Iberdomide; CC-220; Lenalidomide; MM; NDMM; Maintenance; Autologous stem cell transplant; ASCT; CELMoD; Cereblon Modulators
MeSH Terms: conditions — Multiple Myeloma | interventions — iberdomide; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Arm A1: Iberdomide Dose 1 (Experimental)
  Interventions: Drug: Iberdomide
- Arm A2: Iberdomide Dose 2 (Experimental)
  Interventions: Drug: Iberdomide
- Arm A3: Iberdomide Dose 3 (Experimental)
  Interventions: Drug: Iberdomide
- Arm B: Lenalidomide (Active Comparator)
  Interventions: Drug: Lenalidomide

INTERVENTIONS:
Drug: Iberdomide — Specified dose on specified days
  Other Names: CC-220; BMS-986382
  Arms: Arm A1: Iberdomide Dose 1; Arm A2: Iberdomide Dose 2; Arm A3: Iberdomide Dose 3
Drug: Lenalidomide — Specified dose on specified days
  Other Names: Revlimid®
  Arms: Arm B: Lenalidomide

SUMMARY:
The purpose of this study is to compare the effectiveness of iberdomide maintenance to lenalidomide maintenance therapy after autologous stem cell transplantation (ASCT) in participants with newly diagnosed multiple myeloma (NDMM).

ELIGIBILITY:
Inclusion Criteria

* Confirmed diagnosis of symptomatic multiple myeloma (MM).
* Eastern Cooperative Oncology Group performance status (ECOG) score of 0, 1, or 2.
* Received 3 to 6 cycles of an induction therapy that includes a proteasome inhibitor (PI) and immunomodulatory (IMiD) [eg, bortezomib thalidomide and dexamethasone (VTd), lenalidomide, bortezomib and dexamethasone (RVd)] with or without a CD38 monoclonal antibody, daratumumab + bortezomib/thalidomide/dexamethasone [D-VTd] and daratumumab + bortezomib/ lenalidomide/dexamethasone [D-VRd]), or VCd / daratumumab + bortezomib/cyclophosphamide/dexamethasone [D-VCd], and followed by a single or tandem autologous stem cell transplantation (ASCT). Post-stem cell transplant consolidation is permitted.
* Participants within 12 months (single transplant) or 15 months (tandem transplant) from initiation of induction therapy who achieved at least a partial response (PR) after autologous stem cell transplantation (ASCT) with or without consolidation, according to International Myeloma Working Group (IMWG 2016) criteria.

Exclusion Criteria

* Progressive disease or clinical relapse (as defined by IMWG response criteria) following ASCT with or without consolidation or is not responsive to primary therapy.
* Smoldering myeloma, solitary plasmacytoma or nonsecretory myeloma.
* Known central nervous system/meningeal involvement of MM.
* Prior history of malignancies, other than MM, unless the participant has been free of the disease for ≥ 5 years.
* Other protocol-defined Inclusion/Exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1216 (Estimated)
Dates: Start 2023-06-22 (Actual); Primary Completion 2029-03-15 (Estimated); Study Completion 2036-01-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | Up to 6 years

SECONDARY OUTCOMES:
Achieving minimal residual disease (MRD) negativity in participants with complete response (CR) or better at 12 (± 3) months of maintenance treatment | Up to 6 years
Overall Survival | Up to 12 years
Recommended iberdomide dose for Stage 2 | Up to 1 year
Area under the iberdomide plasma concentration-time curve from time zero to tau | Up to 1 year
Area under the iberdomide plasma concentration-time curve within a dosing interval AUC (TAU) | Up to 1 year
Maximum iberdomide concentration (Cmax) | Up to 1 year
Time to maximum iberdomide plasma concentration (Tmax) | Up to 1 year
Number of participants with adverse events (AEs) | Up to 6 years
Progression-free survival on next line of treatment (PFS2) | Up to 6 years
Achieving MRD negativity in participants with CR or better at any time after the date of randomization | Up to 6 years
Conversion from MRD positive to MRD negative in participants with CR or better | Up to 6 years
Achievement of CR or better and maintaining MRD-negative status in 2 bone marrow aspirate assessments that are a minimum of 1 year apart, without any examination showing MRD positive status in between assessments | Up to 6 years
Time to progression (TTP) | Up to 6 years
Time to next treatment (TTNT) | Up to 6 years
Best response achieved prior to progressive disease (PD) | Up to 6 years
Patient-reported health-related quality of life (HRQoL) outcomes and multiple myeloma-related symptoms as measured by the European Organization for Research and Treatment of Cancer [EORTC] Quality of Life C30 questionnaire (QLQ-C30) | Up to 6 years
Patient-reported HRQoL outcomes and multiple myeloma-related symptoms as measured by the EORTC Quality of Life Multiple Myeloma Module (QLQ-MY20) | Up to 6 years

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (285):
- United States (44):
  - Rocky Mountain Cancer Centers, Aurora, Colorado
  - Mayo Clinic Florida, Jacksonville, Florida
  - Tampa General Hospital, Tampa, Florida
  - H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida
  - Cleveland Clinic, Weston, Florida
  - University Cancer Blood Ctr, Athens, Georgia
  - The Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Augusta University - Georgia Cancer Center, Augusta, Georgia
  - The University of Chicago Medical Center - Duchossois Center for Advanced Medicine, Chicago, Illinois
  - University of Kansas Cancer Center - The Richard and Annette Bloch Cancer Care Pavilion, Westwood, Kansas
  - Maryland Oncology Hematology, PA- Clinton, Clinton, Maryland
  - UMass Memorial Medical Center, Worcester, Massachusetts
  - University of Michigan - Rogel Cancer Center, Ann Arbor, Michigan
  - Henry Ford Health System - The Henry Ford Cancer Institute (HFCI) - Detroit, Detroit, Michigan
  - Cancer & Hematology Centers of Western Michigan (CHCWM), Grand Rapids, Michigan
  - Mayo Clinic Cancer Center (MCCC) - Rochester, Rochester, Minnesota
  - Hattiesburg Clinic - Hematology & Oncology, Hattiesburg, Mississippi
  - Morristown Medical Center, Morristown, New Jersey
  - Local Institution - 0328, Brooklyn, New York
  - Perlmutter Cancer Center at NYU Langone Hematology Oncology Associates-Mineola, Mineola, New York
  - NYU Langone Health, New York, New York
  - Columbia University Medical Center - Herbert Irving Pavilion Location, New York, New York
  - Clinical Research Alliance, Westbury, New York
  - Levine Cancer Institute, Charlotte, North Carolina
  - Novant Health Cancer Institute - Elizabeth, Charlotte, North Carolina
  - Duke University Hospital, Durham, North Carolina
  - Novant Health Cancer Institute Hematology - Forsyth, Winston-Salem, North Carolina
  - Wake Forest University Baptist Medical Center (WFUBMC) - Comprehensive Cancer Center, Winston-Salem, North Carolina
  - Oncology Hematology Care, Inc. - Cincinnati - Galbraith Rd, Cincinnati, Ohio
  - Cleveland Clinic - Fairview Hospital - Cancer Center (Moll Cancer Center), Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Midwest Oncology Associates - Kansas City, Kansas, Ohio
  - Cleveland Clinic - Hillcrest Hospital - Hillcrest Cancer Center, Mayfield Heights, Ohio
  - Local Institution - 0013, Toledo, Ohio
  - Wooster Milltown Specialty and Surgery Center, Wooster, Ohio
  - Willamette Valley Cancer Institute, Eugene, Oregon
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center - Jeanes Campus, Philadelphia, Pennsylvania
  - University of Pittsburgh - Hillman Cancer Center, Pittsburgh, Pennsylvania
  - West Cancer Center, Germantown, Tennessee
  - Tennessee Oncology, Nashville, Tennessee
  - Texas Oncology - Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - UT Southwestern-Harold C. Simmons Cancer Center, Dallas, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas
- Argentina (5):
  - Hospital Italiano de Buenos Aires, Ciudad Autonoma Buenos Aires, Buenos Aires F.D.
  - "Centro de Educación Médica e Investigaciones Clínicas ""Norberto Quirno""", Ciudad Autonoma Buenos Aires, Buenos Aires F.D.
  - Local Institution - 0259, Mar del Plata, B
  - Hospital Universitario Austral, Pilar, B
  - Sanatorio Allende, Córdoba
- Australia (4):
  - Calvary Mater Newcastle, Waratah, New South Wales
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Box Hill Hospital, Box Hill, Victoria
  - Monash Health, Clayton, Victoria
- Austria (4):
  - Ordensklinikum Linz Elisabethinen, Linz
  - Universitätsklinikum St. Pölten, Sankt Pölten
  - Medizinische Universitaet Wien - Universitaetsklinik fuer Augenheilkunde und Optometrie, Vienna
  - Hanusch-Krankenhaus, Vienna
- Belgium (2):
  - Grand Hopital de Charleroi - Les Viviers, Charleroi, WHT
  - AZ Groeninge - Campus Kennedylaan, Kortrijk
- Brazil (11):
  - Local Institution - 0245, Curitiba, Paraná
  - CHN - Complexo Hospitalar de Niteroi, Niterói, Rio de Janeiro
  - Instituto Nacional de Câncer, Rio de Janeiro, Rio de Janeiro
  - Hospital das Clínicas da Faculdade de Medicina de Ribeirão Preto da Universidade de São Paulo, Ribeirão Preto, São Paulo
  - Clinica Medica Sao Germano, São Paulo, São Paulo
  - Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo, São Paulo, São Paulo
  - Hospital Santa Marcelina, São Paulo, São Paulo
  - Hospital de Câncer de Barretos - Fundação Pio XII, Barretos
  - Hospital Mãe de Deus, Porto Alegre
  - Instituto COI de Pesquisa, Educação e Gestão, Rio de Janeiro
  - Hospital São Rafael, Salvador
- Canada (4):
  - Cross Cancer Institute, Edmonton, Alberta
  - The Ottawa Hospital - General Campus, Ottawa, Ontario
  - Jewish General Hospital, Montreal, Quebec
  - CHUQ - The Hôtel-Dieu de Québec, Québec, Quebec
- Chile (3):
  - Fundación Arturo López Pérez, Santiago
  - Local Institution - 0258, Temuco
  - Clinica Alemana - Vitacura, Vitacura
- China (37):
  - Anhui Provincial Hospital, Hefei, AH
  - The Fifth Medical Center of People's Liberation Army General Hospital, Beijing, Beijing Municipality
  - Local Institution - 0326, Beijing, BJ
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Local Institution - 0321, Chongqing, CQ
  - Nanfang Hospital of Southern Medical University, Guangzhou, GD
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - Shenzhen Second People's Hospital, Shenzhen, Guangdong
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The Third Xiangya Hospital of Central South University, Changsha, HN
  - Xiangya Hospital, Central South University, Changsha, HN
  - Nanjing Drum Tower Hospital - The Comprehensive Cancer Center, Nanjing, Jiangsu
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - Local Institution - 0263, Nanchang, Jiangxi
  - The First Hospital of Jilin University, Changchun, JL
  - Local Institution - 0094, Shenyang, Liaoning
  - Qilu Hospital of Shandong University, Jinan, SD
  - Xijing Hospital, Xi'an, Shaanxi
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - Local Institution - 0271, Shanghai, Shanghai Municipality
  - Shanghai Fourth People's Hospital, Shanghai, SH
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital - Zhejiang University School of Medicine, Hangzhou, ZJ
  - The First Affiliated Hospital of Ningbo University, Ningbo, ZJ
  - Beijing Chaoyang Hospital, Capital Medical University, Beijing
  - Peking University People's Hospital, Beijing
  - The Second Xiangya Hospital of Central South University, Changsha
  - Fujian Medical University Union Hospital, Fuzhou
  - Sun Yat-sen University Cancer Center, Guangzhou
  - Shandong Provincial Hospital, Jinan
  - Jiangsu Province Hospital, Nanjing
  - Qingdao Municipal Hospital, Qingdao
  - Ruijin Hospital Affiliated to The Shanghai Jiao Tong University Medical School, Shanghai
  - The First Affiliated Hospital of Soochow University, Suzhou
  - Wenzhou Medical University - The First Affiliated Hospital, Wenzhou
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan
  - Tongji Hospital, Tongji Medical College of Huazhong University of Science and Technology, Wuhan
- Colombia (6):
  - Oncomedica S.A., Montería, COR
  - Instituto Nacional de Cancerología - Bogota, Bogotá
  - Fundacion Centro de Tratamiento e Investigacion sobre Cancer Luis Carlos Sarmiento Angulo - CTIC, Bogotá
  - Fundacion Oftalmologica de Santander - FOSCAL, Floridablanca
  - Hospital Pablo Tobon Uribe, Medellín
  - Sociedad de Oncologia y Hematologia del Cesar S.A.S, Valledupar
- Czechia (4):
  - Fakultní Nemocnice Brno, Brno
  - Fakultní Nemocnice Olomouc, Olomouc
  - Fakultní nemocnice Královské Vinohrady, Prague
  - Všeobecná fakultní nemocnice v Praze, Prague
- Odense Universitetshospital, Odense, Denmark
- Finland (2):
  - Helsingin Yliopistollinen Sairaala (HUS) - Syopakeskus (Comprehensive Cancer Center), Helsinki
  - Kuopio University Hospital, Kuopio
- France (10):
  - CHU Hôpital Sud, Amiens
  - Institut d'Hématologie de Basse-Normandie (IHBN), Caen
  - CHU Hôpital Henri Mondor, Créteil
  - Centre Hospitalier Départemental Vendée - Hôpital de la Roche-sur-Yon, La Roche-sur-Yon
  - Centre Hospitalier Régional Universitaire de Lille (CHRU) - Hôpital Claude Huriez, Lille
  - CHU Limoges - Hôpital Dupuytren, Limoges
  - Centre Hospitalier Universitaire de Nantes (CHU de Nantes) - Hotel-Dieu, Nantes
  - Hôpital Saint-Antoine, Paris
  - Hopital Pitie-Salpetriere, Paris
  - Institut Universitaire du Cancer de Toulouse - Oncopole, Toulouse
- Germany (17):
  - Universitätsklinikum Ulm, Ulm, Baden-Wurttemberg
  - Local Institution - 0324, Augsburg, Bavaria
  - Klinikum Bayreuth GmbH, Bayreuth, Bavaria
  - Universitaetsklinikum Erlangen - Medizinische Klinik 5, Erlangen, Bavaria
  - LMU Klinikum der Universitaet Muenchen - Campus Grosshadern - Transplantation, Munich, Bavaria
  - Carl-Thiem-Klinikum Cottbus GmbH, Cottbus, Brandenburg
  - Asklepios Klinik Altona, Hamburg, Hamburg
  - Local Institution - 0313, Hildesheim, Lower Saxony
  - Klinikum Chemnitz gGmbH, Chemnitz, Saxony
  - Charite-Universitaetsmedizin Berlin - Campus Benjamin Franklin (CBF), Berlin, State of Berlin
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - Local Institution - 0310, Göttingen
  - Universitätsklinikum Hamburg-Eppendorf (UKE), Hamburg
  - St. Barbara-Klinik Hamm-Heessen GmbH, Hamm
  - Universitätsklinikum Jena, Jena
  - Local Institution - 0323, Marburg
  - Universitätsklinikum Tübingen, Tübingen
- Greece (6):
  - "General Hospital of Thessaloniki ""G. Papanikolaou""", Thessaloniki, B
  - University of Patras - Rio Regional University Hospital, Rio, G
  - Evangelismos General Hospital of Athens, Athens, I
  - Alexandra General Hospital of Athens, Athens
  - University of Thessaly- General University Hospital of Larissa, Larissa
  - Theageneio Cancer Hospital of Thessaloniki, Thessaloniki
- Queen Mary Hospital, Hong Kong, HK, Hong Kong
- Debreceni Egyetem Klinikai Központ III. sz. Belgyógyászati Klinika, Debrecen, HB, Hungary
- India (10):
  - Postgraduate Institute of Medical Education & Research (PGIMER), Chandigarh, Chandigarh
  - HCG Cancer Center - Kalinga Rao Road, Bangalore, Karnataka
  - Aster Medcity, Kochi, Kerala
  - Dr. Bafnas Star Superspecaility Clinic and Hospital, Kolhāpur, Maharashtra
  - Alexis Multispeciality Hospital, Nagpur, Maharashtra
  - Deenanath Mangeshkar Hospital & Research Center, Pune, Maharashtra
  - Sahyadri Super Speciality Hospital, Pune, Maharashtra
  - Sparsh Hospitals & Critical Care, Bhubaneswar, Odisha
  - Tata Medical Center, Kolkata, West Bengal
  - Local Institution - 0135, Navi Mumbai
- Israel (9):
  - Assuta Medical Center, Ashdod
  - Assaf Harofeh Medical Center, Beer Ya'Aqov
  - Hillel Yaffe Medical Center, Hadera
  - Rambam Medical Center, Haifa
  - Shaare Zedek Medical Center, Jerusalem
  - Hadassah University Medical Center, Jerusalem
  - Rabin Medical Center - Davidoff Center, Petah Tikva
  - The Chaim Sheba Medical Center, Ramat Gan
  - Local Institution - 0136, Tel Aviv
- Italy (11):
  - Azienda Ospedaliero Universitaria Policlinico G. Rodolico San Marco - Ospedale San Marco, Catania, CT
  - Azienda Ospedaliero-Universitaria Careggi, Florence, FI
  - Ospedale Policlinico San Martino, Genova, GE
  - Fondazione IRCCS Cà Granda Ospedale Maggiore Policlinico, Milan, MI
  - ASST Grande Ospedale Metropolitano Niguarda, Milan, MI
  - Azienda Ospedaliero Universitaria Pisana - Ospedale Santa Chiara, Pisa, PI
  - Fondazione Policlinico Universitario Agostino Gemelli, Roma, RM
  - Azienda Ospedaliera Universitaria Citta della Salute e della Scienza di Torino - Ospedale Molinette, Torino, TO
  - "Azienda Ospedaliera Universitaria ""Federico II""", Naples
  - Fondazione IRCCS Policlinico San Matteo, Pavia
  - Policlinico Umberto I, Rome
- Japan (24):
  - National Hospital Organization (NHO) - Shibukawa Medical Center, Shibukawa-shi, Gunma
  - Shonan Kamakura General Hospital, Kamakura-Shi, Kanagawa
  - Kumamoto University Hospital, Kumamoto, Kumamoto
  - Shizuoka Cancer Center, Sunto-gun, Shizuoka
  - Chiba University Hospital, Chiba
  - Gifu Municipal Hospital, Gifu
  - Local Institution - 0133, Higashiibaraki-Gun
  - Hiroshima Red Cross Hospital & Atomic-Bomb Survivors Hospital, Hiroshima
  - Tokai University Hospital, Isehara-shi
  - Nihon University Itabashi Hospital, Itabashi-Ku
  - Kagoshima University Hospital, Kagoshima
  - Kanazawa University Hospital, Kanazawa
  - Local Institution - 0134, Kobe
  - The Cancer Institute Hospital of Japanese Foundation for Cancer Research (JFCR), Kōtoku
  - Gunma University Hospital, Maebashi
  - The Jikei University Hospital, Minatoku
  - The Japanese Red Cross Nagasaki Genbaku Hospital, Nagasaki
  - Nagoya City University Hospital, Nagoya
  - Nerima Hikarigaoka Hospital, Nerima-Ku
  - Jichi Medical University Saitama Medical Center, Saitama-shi
  - Kindai University Hospital, Sakaishi
  - Sapporo Hokuyu Hospital, Sapporo
  - National Hospital Organization Sendai Medical Center, Sendai
  - Japanese Red Cross Medical Center, Shibuya-ku
- Mexico (4):
  - Local Institution - 0127, Mexico City, Mexico City
  - Local Institution - 0283, Monterrey, Nuevo León
  - Phylasis Clinicas Research S.de R.L. de C.V. (PCR)-Toluca, Toluca, State of Mexico
  - Local Institution - 0107, Mexico City
- Netherlands (3):
  - VU University Medical Center, Amsterdam, North Holland
  - Local Institution - 0325, Almere Stad
  - Albert Schweitzer Hospital - Locatie Dordwijk, Dordrecht
- Poland (8):
  - Szpital Uniwersytecki Nr. 2 im Dr. Jana Biziela w Bydgoszczy, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Uniwersyteckie Centrum Kliniczne, Gdansk, Pomeranian Voivodeship
  - Local Institution - 0327, Bydgoszcz
  - Maria Sklodowska-Curie Memorial Cancer Center and Institute of Oncology Gliwice Branch, Gliwice
  - Pratia Onkologia Katowice, Katowice
  - Office of Dr n. Med. Wojciech Legiec, Lublin
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie - Panstwowy Instytut Badawczy, Warsaw
  - Wojewódzkie Wielospecjalistyczne Centrum Onkologii i Traumatologii im. M. Kopernika w Łodzi, Lodz, Łódź Voivodeship
- Portugal (3):
  - Unidade Local de Saude Braga, Braga
  - Unidade Local de Saude de Coimbra, EPE - Hospitais da Universidade de Coimbra, Coimbra
  - Instituto Português Oncologia do Porto Francisco Gentil, EPE, Porto
- Romania (5):
  - Institutul Clinic Fundeni, Bucharest, B
  - Spitalul Clinic Municipal Filantropia Craiova, Craiova, Dolj
  - Institutul Regional de Oncologie Iași, Iași, IS
  - "Institutul Oncologic ""Prof. Dr. Ion Chiricuţă"" Cluj Napoca", Cluj-Napoca, Jud. Cluj
  - "Institutul Oncologic ""Prof. Dr. Ion Chiricuţă"" Cluj Napoca", Cluj-Napoca
- Singapore (2):
  - National University Hospital (S) Pte Ltd, Singapore
  - Singapore General Hospital, Singapore
- South Korea (6):
  - Pusan National University Hospital, Busan
  - National Cancer Center, Goyang-si
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Yonsei University Health System, Severance Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Ulsan University Hospital (UUH), Ulsan
- Spain (10):
  - Hospital Clínic de Barcelona, Barcelona, B
  - Hospital San Pedro de Alcántara, Cáceres, CC
  - Hospital Universitario de Gran Canaria Doctor Negrín, Las Palmas de Gran Canaria, Las Palmas
  - Hospital Universitario Virgen Arrixaca, Murcia, MU
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias
  - Hospital Universitari i Politècnic La Fe, Valencia, VC
  - Hospital Universitari Germans Trias i Pujol, Badalona
  - Clínica Universidad de Navarra -Madrid, Madrid
  - Hospital Universitari Son Espases, Palma de Mallorca
  - Clínica Universidad de Navarra, Pamplona
- Sweden (3):
  - Local Institution - 0171, Luleå, BD
  - Södra Älvsborgs Sjukhus, Borås
  - Vastra Goetalandsregionen - Uddevalla Sjukhus (US), Uddevalla
- Local Institution - 0168, Aarau, Switzerland
- Taiwan (6):
  - E-DA Cancer Hospital, Kaohsiung City
  - Chang Gung Medical Foundation - Kaohsiung Branch, Kaohsiung City
  - Far Eastern Memorial Hospital, New Taipei City
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Chang Gung Memorial Hospital, Taoyuan District
- Turkey (Türkiye) (9):
  - Ankara Bilkent City Hospital, Ankara
  - Liv Hospital Ankara, Çankaya
  - Trakya Üniversitesi Tıp Fakültesi, Edirne
  - Local Institution - 0068, Istanbul
  - T.C. Istanbul Bilim Universitesi - lstanbul Florence Nightingale Hastanesi, Istanbul
  - Ege Universitesi Tip Fakultesi Hastanesi (Ege University Medical Faculty Hospital), Izmir
  - Local Institution - 0073, Izmir
  - Erciyes Üniversitesi Tıp Fakültesi, Kayseri
  - Dr. Abdurrahman Yurtaslan Ankara Onkoloji Eğitim ve Araştırma Hastanesi, Yenimahalle
- United Kingdom (9):
  - NHS Grampian - Aberdeen Royal Infirmary, Aberdeen, ABD
  - GenesisCare -Windosr, Windsor, Berkshire
  - University Hospitals of Derby and Burton NHS Foundation Trust - Royal Derby Hospital, Derby, DBY
  - University Hospitals Dorset NHS Foundation Trust (UHD) - Royal Bournemouth Hospital (RBH), Bournemouth, DOR
  - Portsmouth Hospitals NHS Trust - Queen Alexandra Hospital, Portsmouth, HAM
  - University Hospitals of North Midlands NHS Trust (UHNM) - Royal Stoke University Hospital, Stoke-on-Trent, Staffordshire
  - NHS Lothian - Western General Hospital, Edinburgh
  - Barts Health NHS Trust - St Bartholomew's Hospital, London
  - GenesisCare-Oxford, Oxford

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myer Squibb's data sharing policy and process can be found at https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT05827016.html